CLINICAL TRIAL: NCT04570137
Title: Effects Dietary Fiber From Grains or Fruits and Vegetables on the Intestinal Production of Short-chain Fatty Acids
Brief Title: Fiber Fermentation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hohenheim (Other)
Responsible Party: Principal Investigator, Stephan C. Bischoff, MD, Professor, Prof. Dr., University of Hohenheim
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: FiberStudy
Record Dates: First submitted 2020-09-15; First posted 2020-09-30 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Intestinal Health
Keywords: Gastroenterology; Gut microbiome; Gut barrier

STUDY DESIGN:
Intervention Model Description: Two-armed crossover trial
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): This arm received the arabinoxylan/ß-glucan mix first.
  Interventions: Dietary Supplement: Dietary fiber supplementation
- 2 (Experimental): This arm received the inulin/oligofructose mix first.
  Interventions: Dietary Supplement: Dietary fiber supplementation

INTERVENTIONS:
Dietary Supplement: Dietary fiber supplementation — 1. 16g/day: mix of 70% wheat-bran arabinoxylan and 30% oat-derived fiber (ß-glucan)
  2. 16g/day: mix of 50% inulin and 50% oligofructose from chicory

SUMMARY:
The aim of the study is to better understand the interplay between the intake of dietary fiber and intestinal bacteria, their metabolic activity and the effect on the intestinal barrier.

The effect of two different dietary fiber supplements is tested (arabinoxylan & ß-glucan versus inulin & fructooligosaccharides) in a randomized crossover intervention trial including healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years
* signed written informed consent
* willingness not to change the dietary pattern in the course of the study

Exclusion Criteria:

* BMI below 18 or above 30
* acute or chronic gastrointestinal symptoms
* neoplastic diseases
* very strict diets, including raw foodists and frutarians
* regular smoking (more than one box per day)
* intake of antibiotics, immunosuppressants, or any intestinal therapeutics three months prior to study begin
* supplementation of fibers three months prior to study begin
* simultaneous participation in another clinical study
* pregnancy / breastfeeding
* relevant violations of the study protocol
* intolerance to the fiber supplements (including wheat, oat, chicory)
* occurrence of relevant diseases (individual decision by study physicians)
* revocation of consent
* placement in a clinic or similar facility based on an official or court order

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Short-chain fatty acids (SCFAs) | Will be measured in approx. 4 weeks after study completion.
  SCFAs in native fecal samples

SECONDARY OUTCOMES:
Gut microbiome composition | Will be measured in approx. 6-8 weeks after study completion.
  16S NGS sequencing
Gut barrier integrity | Will be measured in approx. 4 weeks after study completion.
  Lipopolysaccharide-binding protein (plasma) and zonulin (feces)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan C Bischoff, Prof., MD, Principal Investigator — University of Hohenheim, Institute of Nutritional Medicine
Locations (1):
- Institute of Nutritional Medicine, University of Hohenheim, Stuttgart, Germany

IPD SHARING:
Plan to Share IPD: No